CLINICAL TRIAL: NCT00438815
Title: LEVP2006-1 CHANGE 2 Trial (C1-Inhibitor in Hereditary Angioedema Nanofiltration Generation Evaluating Efficacy): Open-Label Safety/Efficacy Repeat Exposure Study of C1INH-nf (Human) in the Treatment of Acute HAE Attacks
Brief Title: Open-Label C1 Esterase Inhibitor (C1INH-nf) for the Treatment of Acute Hereditary Angioedema (HAE) Attacks
Acronym: CHANGE 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEVP2006-1
Record Dates: First submitted 2007-02-21; First posted 2007-02-22 (Estimated); Results first posted 2010-06-09 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Hereditary Angioedema
Keywords: Hereditary angioedema; C1 esterase inhibitor (human)
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — Complement C1 Inhibitor Protein

ARMS (1):
- Open-label C1INH-nf (Experimental): 1,000 Units (U) of C1INH-nf administered intravenously. If there was no response to treatment 60 minutes after the first dose, a second 1,000 U dose could be administered.
  Interventions: Biological: C1 esterase inhibitor [human] (C1INH-nf)

INTERVENTIONS:
Biological: C1 esterase inhibitor [human] (C1INH-nf)

SUMMARY:
The study objective was to evaluate the safety and efficacy of repeat use of C1INH-nf for the treatment of acute HAE attacks.

DETAILED DESCRIPTION:
A total of 113 subjects were enrolled in the study. One-hundred-one (101) subjects received C1INH-nf for the treatment of 1 or more HAE attacks and were analyzed for efficacy. The study design also allowed for short-term prophylaxis with C1INH-nf prior to emergency or non-cosmetic surgical or dental procedures, and an additional 12 subjects received C1INH-nf only for this purpose. All 113 subjects were exposed to C1INH-nf and analyzed for safety.

ELIGIBILITY:
Inclusion Criteria:

This study was open to all subjects who:

* Completed participation in LEVP2005-1/A (NCT00289211) and were not participating in LEVP2005-1/B (NCT01005888), any time after the 3-day telephone follow-up
* Completed participation in LEVP2005-1/B any time after the final prophylactic therapy in Part B
* Were enrolled but not randomized in LEVP2005-1/A after Part A was closed
* Were excluded from LEVP2005-1 for any of the following reasons:

  * Pregnancy or lactation
  * Age less than 6 years
  * Narcotic addiction
  * Presence of anti-C1INH autoantibodies
* Were not enrolled in LEVP2005-1 after enrollment in LEVP2005-1 was closed, under the following circumstances:

  * Had a diagnosis of HAE: evidence of a low C4 level plus either a low C1INH antigenic level or a low C1INH functional level, or
  * Had a known HAE-causing C1INH mutation, or
  * Had a diagnosis of HAE based on a strong family history of HAE as determined by the principal investigator

Exclusion Criteria:

* History of allergic reaction to C1INH or other blood products
* Participated in any other investigational drug study within the past 30 days
* Received blood or a blood product in the past 60 days other than C1INH-nf

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2006-09-21 (Actual); Primary Completion 2009-03-31 (Actual); Study Completion 2009-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (30):
- United States (30):
  - Allergy and Immunology Associates, Scottsdale, Arizona
  - Allergy and Asthma Clinic of Northwest Arkansas, Bentonville, Arkansas
  - UCLA-David Geffen School of Medicine, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - Allergy and Asthma Clinical Research, Inc, Walnut Creek, California
  - Allergy and Asthma Center, Fort Lauderdale, Florida
  - Orlando Regional Healthcare, Orlando, Florida
  - Family Allergy and Asthma Center, Atlanta, Georgia
  - Welborn Clinic Allergy and Immunology, Evansville, Indiana
  - Institute for Asthma and Allergy, Wheaton, Maryland
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Grand Traverse Allergy, Traverse City, Michigan
  - MeritCare Clinical Research, Bemidji, Minnesota
  - Nevada Access to Research and Education Society, Las Vegas, Nevada
  - UMDNJ Asthma and Allergy Research Center, Newark, New Jersey
  - Winthrop University Hospital, Mineola, New York
  - Mount Sinai School of Medicine, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - MeritCare Clinical Research, Fargo, North Dakota
  - Allergy & Asthma Centre of Dayton, Centerville, Ohio
  - Allergy Clinic of Tulsa, Tulsa, Oklahoma
  - Allergy Asthma and Dermatology Research Center, Lake Oswego, Oregon
  - Penn State University, Hershey, Pennsylvania
  - Allergy Partners of the Upstate, Greenville, South Carolina
  - AARA Research Center, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Allergy and Asthma Research Center, San Antonio, Texas
  - Marycliff Allergy Specialists, Spokane, Washington
  - Cornerstone Healthcare, Parkersburg, West Virginia

REFERENCES:
- [Derived] Baker JW, Craig TJ, Riedl MA, Banerji A, Fitts D, Kalfus IN, Uknis ME. Nanofiltered C1 esterase inhibitor (human) for hereditary angioedema attacks in pregnant women. Allergy Asthma Proc. 2013 Mar-Apr;34(2):162-9. doi: 10.2500/aap.2013.34.3645. PMID 23484892
- [Derived] Lumry W, Manning ME, Hurewitz DS, Davis-Lorton M, Fitts D, Kalfus IN, Uknis ME. Nanofiltered C1-esterase inhibitor for the acute management and prevention of hereditary angioedema attacks due to C1-inhibitor deficiency in children. J Pediatr. 2013 May;162(5):1017-22.e1-2. doi: 10.1016/j.jpeds.2012.11.030. Epub 2013 Jan 11. PMID 23312695
- [Derived] Grant JA, White MV, Li HH, Fitts D, Kalfus IN, Uknis ME, Lumry WR. Preprocedural administration of nanofiltered C1 esterase inhibitor to prevent hereditary angioedema attacks. Allergy Asthma Proc. 2012 Jul-Aug;33(4):348-53. doi: 10.2500/aap.2012.33.3585. PMID 22856635
- [Derived] Riedl MA, Hurewitz DS, Levy R, Busse PJ, Fitts D, Kalfus I. Nanofiltered C1 esterase inhibitor (human) for the treatment of acute attacks of hereditary angioedema: an open-label trial. Ann Allergy Asthma Immunol. 2012 Jan;108(1):49-53. doi: 10.1016/j.anai.2011.10.017. Epub 2011 Nov 21. PMID 22192966
- [Derived] Zuraw BL, Busse PJ, White M, Jacobs J, Lumry W, Baker J, Craig T, Grant JA, Hurewitz D, Bielory L, Cartwright WE, Koleilat M, Ryan W, Schaefer O, Manning M, Patel P, Bernstein JA, Friedman RA, Wilkinson R, Tanner D, Kohler G, Gunther G, Levy R, McClellan J, Redhead J, Guss D, Heyman E, Blumenstein BA, Kalfus I, Frank MM. Nanofiltered C1 inhibitor concentrate for treatment of hereditary angioedema. N Engl J Med. 2010 Aug 5;363(6):513-22. doi: 10.1056/NEJMoa0805538. PMID 20818886

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-label C1INH-nf: 1,000 Units (U) of C1 esterase inhibitor (C1INH-nf) administered intravenously (IV). If there was no response to treatment 60 minutes after the first dose, a second 1,000 U dose could be administered.
Period: Overall Study
Arm/Group | Open-label C1INH-nf
Started | 113
Completed | 43
Not Completed | 70
Not completed — Transferred to LEVP2006-4 (NCT00462709) | 30
Not completed — 3-month follow-up no longer required | 12
Not completed — Noncompliance with protocol requirements | 9
Not completed — Transitioned to commercial C1INH-nf | 6
Not completed — Lost to Follow-up | 6
Not completed — Withdrawal by Subject | 6
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Groups:
- Open-label C1INH-nf: 1,000 U of C1INH-nf administered IV. If there was no response to treatment 60 minutes after the first dose, a second 1,000 U dose could be administered.
Arm/Group | Open-label C1INH-nf
Number analyzed (Participants) | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (17.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75
  Male | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Hereditary Angioedema (HAE) Attacks Treated With C1INH-nf
Time Frame: Duration of the study (2.5 years)
Population: Intent-to-treat Efficacy (ITT-E) Population (N=101; the number of subjects who received at least one dose of C1INH-nf for the treatment of an acute HAE attack).
Measure: Number; unit: attacks
Arm/Group | Open-label C1INH-nf
Number analyzed (Participants) | 101
attacks
  Conservative Analysis | 609
  Less Conservative Analysis | 598

2. Secondary Outcome: Time to Beginning of Substantial Relief of the Defining Symptom
Description: Subjects were to assess their symptoms every 15 minutes up to 4 hours after the initial dose or until substantial relief of the defining symptom was achieved. Substantial relief was defined as 3 consecutive assessments of improvement of the defining symptom. Beginning of substantial relief was considered the first of the 3 consecutive assessments.
Time Frame: Within 4 hours after initial treatment
Population: ITT-E Population.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Open-label C1INH-nf
Number analyzed (Participants) | 101
hours | 0.75 [0.50 to 1.00]

3. Secondary Outcome: Time to Beginning of Substantial Relief of the Defining Symptom for Subjects Who Received Multiple Treatments
Description: For attack number 1, the number of censored observations precluded estimation of the 95% confidence interval (CI) upper bound for median time to event (subjects who did not experience beginning of substantial relief of the defining symptom within 4 hours after initial treatment were included in the analysis as censored observations). Entry of 4.0 hours indicates that data were not estimable (NE); as non-numeric data are not supported by the 95% CI field, entry of the actual result (ie, NE or >4.0) was not possible.
Time Frame: Within 4 hours after initial treatment
Population: ITT-E subjects with at least 10 HAE attacks during the study (N=15).
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Open-label C1INH-nf
Number analyzed (Participants) | 15
hours
  Attack number 1 | 1.50 [0.75 to 4.00]
  Attack number 2 | 0.50 [0.25 to 2.50]
  Attack number 3 | 0.50 [0.50 to 0.75]
  Attack number 4 | 0.50 [0.25 to 1.00]
  Attack number 5 | 0.75 [0.50 to 1.25]
  Attack number 6 | 0.50 [0.25 to 1.25]
  Attack number 7 | 0.75 [0.50 to 0.75]
  Attack number 8 | 0.50 [0.25 to 0.75]
  Attack number 9 | 0.25 [0.25 to 0.50]
  Attack number 10 | 0.50 [0.25 to 0.75]

4. Secondary Outcome: Antigenic C1 Inhibitor (C1INH) Serum Levels
Description: Change in antigenic C1INH serum levels from pre-infusion to 1 hour after the initial dose of study drug.
Time Frame: Pre-infusion to 1 hour post-infusion
Population: ITT-E subjects with data at both sampling time points (N=84).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Open-label C1INH-nf
Number analyzed (Participants) | 84
mg/dL
  Pre-infusion | 10.7 (13.91)
  Increase at 1 hour post-infusion | 9.6 (12.98)

5. Secondary Outcome: Functional C1INH Serum Levels
Description: Percent change in functional C1INH serum levels from pre-infusion to 1 hour after the initial dose of study drug. Functional C1INH serum levels are expressed as a percent of total detectable C1INH (ie, functional C1INH/total detectable C1INH).
Time Frame: Pre-infusion to 1 hour post-infusion
Population: ITT-E subjects with data at both sampling time points (N=82).
Measure: Mean (Standard Deviation); unit: percent of functional C1INH
Arm/Group | Open-label C1INH-nf
Number analyzed (Participants) | 82
percent of functional C1INH
  Pre-infusion | 27.0 (19.30)
  Percent increase at 1 hour post-infusion | 39.2 (18.04)

6. Secondary Outcome: Complement C4 Serum Levels
Description: Change in complement C4 serum levels from pre-infusion to 1 hour after the initial dose of study drug.
Time Frame: Pre-infusion to 1 hour post-infusion
Population: ITT-E subjects with data at both sampling time points (N=74).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Open-label C1INH-nf
Number analyzed (Participants) | 74
mg/dL
  Pre-infusion | 5.3 (5.41)
  Change at 1 hour post-infusion | -0.2 (1.51)

7. Primary Outcome: Percent of HAE Attacks With Substantial Relief of the Defining Symptom
Description: Subjects were to assess their symptoms every 15 minutes up to 4 hours after the initial dose or until substantial relief of the defining symptom was achieved. The conservative analysis defined substantial relief as 3 consecutive assessments of improvement of the defining symptom; any attack that did not have 3 consecutive documented reports of improvement was considered a treatment failure. In the less conservative analysis, attacks also were considered to have responded if clinical improvement of the defining symptom occurred but data were incomplete due to cessation of symptom assessments.
Time Frame: Within 4 hours after initial treatment
Population: ITT-E Population (N=101; the number of subjects who received at least one dose of C1INH-nf for the treatment of an acute HAE attack).
Measure: Number; unit: percent of attacks
Arm/Group | Open-label C1INH-nf
Number analyzed (Participants) | 101
percent of attacks
  Conservative Analysis | 87
  Less Conservative Analysis | 95

ADVERSE EVENTS:
Description: Presented are all treatment-emergent adverse reactions considered to be related to C1INH-nf.
Arm/Group | Open-label C1INH-nf
Serious Adverse Events (participants affected / at risk) | 0/113
Other Adverse Events (participants affected / at risk) | 1/113
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label C1INH-nf (N=113)
Infusion site pain (General disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement. Most restrictive provision - PI will not publish results until after first of: multicenter publication is published or 24 months from study end. Thereafter, PI may publish his results. PI must provide copy of proposed publication to sponsor for pre-review. If sponsor requests, PI must delete sponsor confidential information before publication and/or delay publication for 90 days so sponsor can file for patents or take other action to protect its patent rights.